CLINICAL TRIAL: NCT04628364
Title: A Systems-based Approach to Patient-focused Rare Disease Research and Product Development
Brief Title: The Natural History of Metachromatic Leukodystrophy Study (HOME Study)
Status: Completed | Type: Observational
Sponsor: National Organization for Rare Disorders (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Aliza Fink, Director of Research Programs, National Organization for Rare Disorders
Other Study IDs: 75F40119C10091
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Metachromatic Leukodystrophy
Keywords: MLD; Leukodystrophy; Rare Disease; Natural History Study
MeSH Terms: conditions — Leukodystrophy, Metachromatic; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aims of the HOME Study are to:

* Design and implement a natural history study for metachromatic leukodystrophy to serve as a source of external control data, to augment or replace concurrent controls in clinical trials;
* Pilot test and develop guidance on how to design, conduct, and analyze the data from a natural history study to support adaptive trial designs for regulatory use;
* Reduce burden of participation in trials and provide a potential solution to patient recruitment challenges, particularly for RCT's; and
* Design approaches that support remote participation in studies.

DETAILED DESCRIPTION:
The HOME Study is a web-based natural history study for patients with metachromatic leukodystrophy. It is hosted by the National Organization for Rare Disorders (NORD); an independent non-profit patient advocacy organization dedicated to individuals with rare diseases and the organizations who serve them.

The study collects information from participants (or their authorized respondents, heretofore referred to collectively as "participants") who are affected by metachromatic leukodystrophy.

Data are collected at pre-baseline, baseline, 3, 6, 9, and 12 months through online surveys, telephone Interviews, web-based virtual assessments with a clinical study coordinator, and a (optional - only for U.S. residents) mobile application. Data entered into this study includes name, date of birth, diagnosis, treatments, medical history, family history, quality of life, disease progression, treatment - past and proposed, general medical information, genetic test results and mutations, blood level results, upload of medical records.

ELIGIBILITY:
Inclusion Criteria:

The study is open to English speaking individuals of all ages who have a diagnosis consistent with metachromatic leukodystrophy (MLD). MLD is defined as:

* Mutations in the ASA and PSAP genes identified by genetic testing;
* A diagnosis of MLD by MRI of the brain; or
* Sulfatase enzyme activity and urinary sulfatide excretion identified by biochemical testing.

Exclusion Criteria:

Patients will be excluded from the study if they do not meet inclusion criteria.

* Non-English speaking individuals
* No confirmed diagnosis of metachromatic leukodystrophy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is open to English speaking individuals of all ages who have a diagnosis consistent with metachromatic leukodystrophy (MLD). MLD is defined as:
  * Mutations in the ASA and PSAP genes identified by genetic testing;
  * A diagnosis of MLD by MRI of the brain; or
  * Sulfatase enzyme activity and urinary sulfatide excretion identified by biochemical testing.
  This diagnosis will be confirmed by participant upload of confirmatory test (genetic, blood, urine).
  Participants providing data must be at least 18 years of age, or legally authorized to provide information on behalf of a minor or someone who is unable to provide information themselves. Consent from a legally authorized representative is required for participants who are minors or who are over the age of 18 but unable to provide informed consent. Consent of one parent or legally authorized representative is considered sufficient for participation of a minor in this study and assent will not be collected.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Classification System - Metachromatic Leukodystrophy (GMFC-MLD) | Baseline, 3, 6, 9, 12 months
  The GMFC-MLD consists of seven levels and is applicable from the age of 18 months. It represents all clinically relevant stages from normal (level 0) to loss of all gross motor function (level 6).

SECONDARY OUTCOMES:
Change in Expressive Language Function Classification - Metachromatic Leukodystrophy (ELFC-MLD) | Baseline, 3, 6, 9, 12 months
  Describes expressive language.
Change in WHO Motor Milestone | Baseline, 3, 6, 9, 12 months
  Assessment of six milestones that are fundamental to acquiring self-sufficient, erect locomotion.

CONTACTS AND LOCATIONS:
Locations (1):
- National Organization for Rare Disorders, Danbury, Connecticut, United States

REFERENCES:
- See also: HOME Study overview and enrollment — https://rarediseases.org/mld-home-study/